CLINICAL TRIAL: NCT06156891
Title: Selective De-escalation of Radiotherapy Density Based on Response to Induction Chemotherapy With PD-1 Inhibitor Toripalimab, Docetaxel, Cisplatin, and Capecitabine in Locally Advanced Oropharyngeal Carcinoma: A Prospective Phase II Trial (DEDICATE-1)
Brief Title: PD-1 Inhibitor Based Induction Chemotherapy Followed by De-escalation Protocols in OPSCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoshen Wang, Professor, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022145-1
Record Dates: First submitted 2023-11-26; First posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Oropharyngeal Cancer
Keywords: Oropharyngeal Cancer; Immune Checkpoint Inhibitor; Induction chemotherapy; De-escalation; HPV-related; HPV-unrelated
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toxicities reduced treatment arm (Experimental): Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) and omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 70% Partial Response(PR) in HPV-related patients.
  Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) combined with concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 70% Partial Response(PR) in HPV-urelated patients.
  Interventions: Procedure: Toxicities reduced treatment
- Conventional treatment arm (Active Comparator): Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by concurrent cisplatin chemoradiotherapy with standard radiation dose (70.4Gy/32Fx) when responses to induction chemotherapy are less than 70% Partial Response (PR) regardless of HPV status.
  Interventions: Procedure: Conventional treatment

INTERVENTIONS:
Procedure: Toxicities reduced treatment — Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) and omitting concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 70% Partial Response(PR) in HPV-related patients.
  Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by reducing radiation dose(60Gy/30Fx) combined with concurrent cisplatin chemotherapy when responses to induction chemotherapy are ≥ 70% Partial Response(PR) in HPV-urelated patients.
  Arms: Toxicities reduced treatment arm
Procedure: Conventional treatment — Two cycles toripalimab+docetaxel+cisplatin+capecitabine (TPF) induction chemotherapy followed by concurrent cisplatin chemoradiotherapy with standard radiation dose (70.4Gy/32Fx) when responses to induction chemotherapy are less than 70% Partial Response (PR) regardless of HPV status.
  Arms: Conventional treatment arm

SUMMARY:
More and more studies have shown that the efficacy and prognosis of HPV （Human papillomavirus）-positive oropharyngeal cancer (OPC) patients are better than those of others. However, in the NCCN (National Comprehensive Cancer Network) Oncology Clinical Guidelines for OPC treatment, each group of p16+ is consistent with the corresponding group of p16-, which indicates that the treatment of OPC is basically the same regardless of whether it is related to HPV. Several studies attempted to reduce the toxicities of treatment of HPV related OPC through reduced-dose radiation and showed promising results, and all of the studies have shown that induction chemotherapy is a good way to screen followed treatment. Those who are effective in induction chemotherapy are usually more sensitive to radiation therapy, and reducing the intensity of subsequent treatment will not affect the survival outcome of patients. Immune checkpoint inhibitors (ICIs) have proved to improve outcomes of head and neck cancers. However, In KEYMAT-048, a Phase III controlled trial of relapsed/metastatic head and neck squamous cell carcinoma, ICIs showed an overall survival advantage, but the survival advantage was independent of HPV status. Therefore, patients with HPV-negative OPC still have a good response to ICIs. So we added anti-PD-1 antibody Toripalimab to induction chemotherapy in order to achieve better response rates to receive de-escalation chemoradiotherapy followed regardless of whether it is related to HPV.

ELIGIBILITY:
Inclusion Criteria:

Histological diagnosis of squamous cell carcinoma of oropharynx; IHC p16 positive or PCR HPV16 positive; IHC p16 negative or PCR HPV16 negative; T3-4N0-3M0 or T1-2N2-3M0 according to UICC/AJCC 8th staging system; Age ≥18; No prior anti-tumor treatment; Informed consent obtained; Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1; Normal complete blood count; Normal hepatic function; Normal renal function (creatinine ≤ 1.5 times the upper limit of normal). -

Exclusion Criteria:

Previous radiotherapy; A history of any other type of malignancy; Pregnancy or lactation; Obvious disfunction of liver, renal, cardiac or lung function; Un controlled infection; Systemic metastasis or distant metastasis; Patients with severe gastrointestinal diseases; Patients with mental disorders affecting patient participation in trial judgement.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 year
  Objective Response Rate
LRRR | 2 year
  locoregional recurrence rate
PFS | 2 year
  progression free survival
OS | 2 year
  overall survival

SECONDARY OUTCOMES:
The percentage of Grade 3 and 4 adverse reactions in NCI-CTC AE 5.0 and RTOG | 2 year
  The incidence (percentage) of late toxicity , Grade 3 and 4 adverse reactions in NCI-CTC AE 5.0 and RTOG.
QoL | 2 year
  Quality of Life according to EORTC QLQ-C30
Number and percentage of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and RTOG | 2 years
  The detail number and percentage of adverse events by every systems Assessed by CTCAE v5.0 and RTOG.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China